CLINICAL TRIAL: NCT01027234
Title: A Phase I, Single-center, Randomized, Double-blind, Placebo-controlled Single-ascending Dose, First Time Into Man Study to Assess the Safety, Tolerability, and Pharmacokinetics (Part A) and an Open-label Assessment of the Effect of Food on the Pharmacokinetics (Part B) of Orally Administered AZD8418
Brief Title: This Study Will Assess the Safety and Tolerability of AZD8418 After Single Increasing Oral Doses
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Pre-Clinical Safety Tox Findings
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: D2590C00001
Record Dates: First submitted 2009-12-04; First posted 2009-12-07 (Estimated); Last update posted 2010-05-26 (Estimated); Status verified 2010-05

CONDITIONS: Healthy
Keywords: Healthy volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: AZD8418
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD8418 — Single oral dose
  Arms: 1
Drug: Placebo — single oral dose
  Arms: 2

SUMMARY:
The main purpose of this study is to assess the safety and tolerability of AZD8418 after single increasing oral doses.

Another purpose of this study is to evaluate the pharmacokinetics (also called PK - how the study drug enters and leaves the body and how your body acts on the study drug) of AZD8418. Part B of the study will assess the effect of food on the safety and pharmacokinetics of AZD8418.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers
* Healthy female volunteers of non-childbearing potential

Exclusion Criteria:

* History of any clinically significant medical, neurologic, or psychiatric disease (including repeated episodes of major depression) or a disorder which, in the opinion of the Investigator, may either put the volunteer at risk because of participation
* History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the Investigator, or history of hypersensitivity to drugs with a similar chemical structure or class to AZD8418

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2009-11; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of AZD8418 following the oral administration of single ascending doses and to estimate the maximum tolerated dose in healthy volunteers. | Safety assessments will be obtained daily throughout the study

SECONDARY OUTCOMES:
To characterise the pharmacokinetics of AZD8418 and its metabolites in plasma and urine, and provisionally assess the dose proportionality of the pharmacokinetics following administration of single ascending doses of AZD8418. | samples will be obtained pre and post dose
To assess the effect of food on the safety and pharmacokinetic profile of AZD8418 and its metabolites. | samples will be obtained pre and post dose

CONTACTS AND LOCATIONS:
Overall Officials: Philip T. Leese, M.D., Principal Investigator — Quintiles, Inc.
Locations (1):
- Research Site, Overland Park, Kansas, United States